CLINICAL TRIAL: NCT02258646
Title: Long-Term Integrated Telerehabilitation of COPD Patients. A Multi-Center Randomized Controlled Trial
Brief Title: Long-Term Integrated Telerehabilitation of COPD Patients. A Multi-Center Trial
Acronym: iTrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Research Council of Norway (Other); The Royal Norwegian Ministry of Health (Other); LHL Helse (Other); University of Tromso (Other); La Trobe University (Other); The Alfred (Other); Aalborg University (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Esbjerg Municipality (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 228919/DHE; HST1117-13 (Other Grant/Funding Number: Northern Norway Regional Health Authority); HST1118-13 (Other Grant/Funding Number: Northern Norway Regional Health Authority)
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Exercise; Rehabilitation; Telemedicine; Treatment Outcome; Costs and Cost Analysis; Physical Therapists; Adaptation, Psychological
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Telerehabilitation (Experimental): Exercise training at home, telemonitoring, and education/self-management
  Interventions: Behavioral: Exercise training at home; Behavioral: Telemonitoring and education/self-management
- Unsupervised exercise training at home (Experimental): Unsupervised exercise training at home
  Interventions: Behavioral: Exercise training at home
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Exercise training at home
  Arms: Telerehabilitation; Unsupervised exercise training at home
Behavioral: Telemonitoring and education/self-management
  Arms: Telerehabilitation

SUMMARY:
This research project aims to conduct a three-arm multi-center randomized controlled trial (RCT) on an innovative telerehabilitation intervention for patients with chronic obstructive pulmonary disease (COPD). The overall purpose of the RCT is to demonstrate whether long-term integrated telerehabilitation involving exercise training at home, telemonitoring, and education/self-management will prevent hospital readmissions, thus reducing healthcare costs, for patients with COPD, and will improve patient status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* At least one COPD-related hospitalization or COPD-related emergency department presentation in the previous 12 months to enrollment
* Capable to provide signed written informed consent

Exclusion Criteria:

* Attendance to a rehabilitation program in the previous 6 months of enrollment
* Participation in another study that may have an impact on the outcome of this study
* Deemed by the health care team to be physically uncapable to perform the study procedures
* Presence of comorbidities wich might prevent the patient from safely undertake an exercise program at home
* Home environment not suitable for installation and use of rehabilitation and monitoring equipment (e.g. physical space, Wi-FI Internet or mobile Internet via 4G)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Combined number of hospitalizations and emergency department presentations | Two years

SECONDARY OUTCOMES:
Hospitalizations | Two years
Emergency department presentations | Two years
Mortality | Two years
Time free from first hospitalization or emergency department presentation | Two years
Cost-effectiveness | Two years
  Cost-Utility Analysis (Cost/QALY)
Change from baseline in COPD Assessment Test at 6 months | 6 months
Change from baseline in COPD Assessment Test at 1 year | One year
Change from baseline in COPD Assessment Test at 2 years | Two years
Change from baseline in EQ-5D at 6 months | Six months
Change from baseline in EQ-5D at 1 year | One year
Change from baseline in EQ-5D at 2 years | Two years
Change from baseline in Hospital Anxiety and Depression Scale at 6 months | Six months
Change from baseline in Hospital Anxiety and Depression Scale at 1 year | One Year
Change from baseline in Hospital Anxiety and Depression Scale at 2 years | Two years
Change from baseline in Generalized Self-Efficacy Scale at 6 months | Six months
Change from baseline in Generalized Self-Efficacy Scale at 1 year | One year
Change from baseline in Generalized Self-Efficacy Scale at 2 years | Two years
Change from baseline in 6- minute walking distance at 6 months | Six months
Change from baseline in 6- minute walking distance at 1 year | One year
Change from baseline in 6- minute walking distance at 2 years | Two years
Change from baseline in physical activity at 6 months | Six months
Change from baseline in physical activity at 1 year | One year
Change from baseline in physical activity at 2 years | Two years
Patient Global Impression of Change after 2 years | Two years
Hospitalizations at 1 year | One year
Emergency department presentations at 1 year | One year
Mortality at 1 year | One year

OTHER OUTCOMES:
Change from baseline in BODE Index at 6 months | 6 months
Change from baseline in BODE Index at 1 year | 1 year
Change from baseline in BODE Index at 2 years | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Zanaboni, PhD, Principal Investigator — University Hospital of North Norway; Anne E Holland, PhD, Principal Investigator — La Trobe University; Birthe Dinesen, PhD, Principal Investigator — Aalborg University
Locations (3):
- The Alfred, Melbourne, Victoria, Australia
- Sydvestjysk Hospital, Esbjerg, Denmark
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Derived] Hoaas H, Zanaboni P, Hjalmarsen A, Morseth B, Dinesen B, Burge AT, Cox NS, Holland AE. Seasonal variations in objectively assessed physical activity among people with COPD in two Nordic countries and Australia: a cross-sectional study. Int J Chron Obstruct Pulmon Dis. 2019 Jun 5;14:1219-1228. doi: 10.2147/COPD.S194622. eCollection 2019. PMID 31239657
- [Derived] Zanaboni P, Dinesen B, Hjalmarsen A, Hoaas H, Holland AE, Oliveira CC, Wootton R. Long-term integrated telerehabilitation of COPD Patients: a multicentre randomised controlled trial (iTrain). BMC Pulm Med. 2016 Aug 22;16(1):126. doi: 10.1186/s12890-016-0288-z. PMID 27549782
- See also: Study website — https://ehealthresearch.no/en/projects/itrain-study